CLINICAL TRIAL: NCT05233891
Title: Validation of Scales in Reconstructive Breast Surgery
Acronym: ValPlast
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-03165
Record Dates: First submitted 2022-01-23; First posted 2022-02-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Hypertrophy
Keywords: plastic surgery; breast reconstruction; patient reported outcome; complication
MeSH Terms: conditions — Breast Neoplasms; Gigantomastia | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast reconstruction after breast cancer: Women who have had/have breast cancer and will have/have had a breast reconstruction.
  Interventions: Procedure: Breast reconstruction
- Breast reduction: Women who have had/will have a breast reduction due to breast hypertrophy.
  Interventions: Procedure: Breast reduction

INTERVENTIONS:
Procedure: Breast reconstruction — Breast reconstruction after breast cancer.
  Groups: Breast reconstruction after breast cancer
Procedure: Breast reduction — Breast reduction due to breast hypertrophy.
  Other Names: mammoplasty reduction
  Groups: Breast reduction

SUMMARY:
The main purpose of the project is to validate patient reported outcomes measures (PROMs) in reconstructive breast surgery. BREAST-Q will be evaluated for Swedish and Sweden.Hospital Anxiety and Depression Scale (HADS), EuroQol 5D (EQ5D), and SF-36 will be validated for reconstructive breast surgery. In addition, the complication classification system according to Clavien-Dindo will be validated for reconstructive breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had or will have reconstructive breast surgery in Sahlgrenska university hospital.

Exclusion Criteria:

* Do not understand Swedish.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are biological women and identify as cis-women.
Study Population: Women who will have or have had reconstructive breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2027-12-21 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Validation and reliability of BREAST-Q for Sweden | Pre-operatively
  Breast-Q measures breast related quality of life on a scale 1-100. A higher score indicates a higher quality of life.
Validation and reliability of BREAST-Q for Sweden | 5 years postoperatively
  Breast-Q measures breast related quality of life on a scale 1-100. A higher score indicates a higher quality of life.
Validation and reliability of EuroQol-5 dimensions, 3 levels for reconstructive breast surgery | Pre-operatively
  EuroQol-5 dimensions-3 levels (EQ5D) is a generic instrument developed for health economic and clinical evaluation of healthcare. A total score between 0 and 1 is calculated. Zero equals death and 1 perfect health.
Validation and reliability of EuroQol-5 dimensions, 3 levels for reconstructive breast surgery | 5 years postoperatively
  EuroQol-5 dimensions-3 levels (EQ5D) is a generic instrument developed for health economic and clinical evaluation of healthcare. A total score between 0 and 1 is calculated. Zero equals death and 1 perfect health.
Validation and reliability of Hospital Anxiety and Depression scale (HADS) for Reconstructive breast surgery | Pre-operatively
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Validation and reliability of Hospital Anxiety and Depression scale (HADS) for Reconstructive breast surgery | 5 years postoperatively
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Validation and reliability of RAND-36 for reconstructive breast surgery | Pre-operatively
  It comprises eight subdomains: physical functioning (10 items), role limitations caused by physical health problems (4 items), role limitations caused by emotional problems (3 items), social functioning (2 items), emotional well-being (5 items), energy/fatigue (4 items), pain (2 items), and general health perceptions (5 items) where patients score their health during the last four weeks on Likert scales. Every item score is transformed linearly to the per cent of total possible score (0-100) and then averaged by the values of the scale. A subscore is calculated for each domain and in addition two summary scores, physical and mental health, are calculated.
Validation and reliability of RAND-36 for reconstructive breast surgery | 5 years postoperatively
  It comprises eight subdomains: physical functioning (10 items), role limitations caused by physical health problems (4 items), role limitations caused by emotional problems (3 items), social functioning (2 items), emotional well-being (5 items), energy/fatigue (4 items), pain (2 items), and general health perceptions (5 items) where patients score their health during the last four weeks on Likert scales. Every item score is transformed linearly to the per cent of total possible score (0-100) and then averaged by the values of the scale. A subscore is calculated for each domain and in addition two summary scores, physical and mental health, are calculated.
Validation of Clavion-Dindo classification for reconstructive breast surgery | 5 years postoperatively
  The Clavien-Dindo system is based on ranking the severity of the intervention required to treat a given complication, as follows: grade I includes deviations from the postoperative course without the need for pharmacological treatment or surgical/endoscopic/radiological intervention; grade II complications require pharmacological treatment, blood transfusion, or total parental nutrition; grade III complications require surgical/endoscopic/radiological intervention; grade IV includes life-threatening complications, including those involving the central nervous system, that require intensive care treatment; and grade V includes complications that result in death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weick L, Brorson F, Jepsen C, Liden M, Jensen EW, Hansson E. Giving meaning to patient reported outcomes in breast reconstruction after mastectomy - A systematic review of available scores and suggestions for further research. Breast. 2022 Feb;61:91-97. doi: 10.1016/j.breast.2021.11.008. Epub 2021 Nov 25. PMID 34929423
- [Result] Kamya L, Hansson E, Weick L, Hansson E. Validation and reliability testing of the Breast-Q latissimus dorsi questionnaire: cross-cultural adaptation and psychometric properties in a Swedish population. Health Qual Life Outcomes. 2021 Jul 3;19(1):174. doi: 10.1186/s12955-021-01812-x. PMID 34217326
- [Result] Weick L, Grimby-Ekman A, Lunde C, Hansson E. Validation and reliability testing of the BREAST-Q expectations questionnaire in Swedish. J Plast Surg Hand Surg. 2023 Feb-Dec;57(1-6):315-323. doi: 10.1080/2000656X.2022.2070180. Epub 2022 May 9. PMID 35533094
- [Derived] Jepsen C, Paganini A, Hansson E. Validation and reliability testing of the Swedish version of the BREAST-Q reconstruction. Scand J Surg. 2025 Oct 26:14574969251387498. doi: 10.1177/14574969251387498. Online ahead of print. PMID 41139858
- See also: Full text article — https://pubmed.ncbi.nlm.nih.gov/35533094/
- See also: Full text article — https://pubmed.ncbi.nlm.nih.gov/34217326/
- See also: Full text article — https://pubmed.ncbi.nlm.nih.gov/34929423/